CLINICAL TRIAL: NCT00990743
Title: Phase I Study With SYL040012. Tolerance and Effect on Intraocular Pressure
Brief Title: Tolerance and Effect on Intraocular Pressure After Administration of SYL040012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Ana Isabel Jiménez, Sylentis
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-008204-41; CUNFI-0511-0814
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Ocular Hypertension; Glaucoma
Keywords: Ocular hypertension; Glaucoma; Beta-blocker
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SYL040012 (Experimental)
  Interventions: Drug: SYL040012

INTERVENTIONS:
Drug: SYL040012 — Administration of single and multiple doses of SYL040012 in ophthalmic drops solution

SUMMARY:
The purpose of this study is to determine whether SYL040012 is safe for the treatment of ocular hypertension and glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, any gender
* 18 to 45 years of age,
* Subjects must provide signed informed consent prior to participation in any study-related procedures
* Body Mass Index between 19,5 and 29 kg/m2
* IOP </= 21 mmHg in both eyes
* Have a BCVA (Best corrected visual acuity) of >/= 0.8 (20/25) (Snellen scale), or </= 0.1 (LogMar units)in both eyes
* Normal Fluorescein Clearance Test in both eyes
* Normal funduscopy in both eyes

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test. Females of childbearing potential who will not use a medically acceptable contraceptive method from selection and during the hole study.
* Current relevant disease, including respiratory disease, cardiovascular, endocrine, neurological, haematological, renal, neoplastic, hepatopathy, gastrointestinal distress, hypertension, or infectious acute processes
* Previous chronic processes or with rebound characteristics that could interfere with study according to the investigator's judgment.
* Volunteers who have received pharmacological treatment, including medicinal plants, during the four weeks previous to beginning the study.
* Having used anti-cholinergics, betablockers and corticoids sporadically in the last 30 days whichever the route of administration, or any med by ocular or nasal administration route.
* Case history of hypersensitivity to meds or any other allergic process
* Visual alterations: Previous eye surgery, glaucoma, uveitis or ocular surface pathology (dry eye, blepharitis).
* Volunteers with visual alteration with more than 3 dioptres in either eye
* Use of contact lenses
* Volunteer who has participated in a clinical trial during the past four months before study entry.
* Blood or derivate transfusion during the six previous months to study entry
* Case history of drug or alcohol abuse or dependence.
* Positive result in test drug abuse during selection period
* Positive serology results to hepatitis B virus (HbsAg), virus C or HIV
* Analytic alterations medically relevant, at investigator's judgement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Part I: Local tolerance after administration of one dose of SYL040012. | Part I: 3 days
Part II: Local tolerance after 7 days administration of SYL040012 with one dose per day. | Part II: 11 days

SECONDARY OUTCOMES:
Period I: Local Tolerance Assessment, Effect Assessment & Pharmacokinetic description after administration of one dose of SYL040012.Side effects. Analytics. | Part I: 1 hour, 1, 2, 3, days
Period II:Tolerance assessment, Pharmacokinetic description, Effect assessment on the IOP after 7 days administration. Side effects. Analytics | Part II: After each administration, at time 1 and 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Belen Sadaba, MD, PhD, Principal Investigator — Clínica Universitaria de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain